CLINICAL TRIAL: NCT05771064
Title: Promoting In-Home Activities at a Memory & Aging Clinic (Pro-Home MeC)
Brief Title: Promoting In-Home Activities at a Memory & Aging Clinic
Acronym: Pro-Home MeC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Naoko Muramatsu, Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2022-1412
Record Dates: First submitted 2022-11-03; First posted 2023-03-16 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: MCI; Mild Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Gentle Moves (Experimental): Three-month physical activity intervention.
  Interventions: Behavioral: Gentle Moves
- Usual Care (No Intervention): Usual care provided by neuropsychologist.

INTERVENTIONS:
Behavioral: Gentle Moves — A safe physical activity program which consists of a brief motivational enhancement and three movements to be performed in a seated position; and two movements in the standing position. The intervention will be delivered by a research coach.
  Arms: Gentle Moves

SUMMARY:
The objective of the proposed study, "Promoting In-Home Activities at a Memory & Aging Clinic (Pro-Home MeC)", is to assess and improve the feasibility of a physical activity (PA) intervention and the measurement of cognitive outcomes in a memory clinic setting for inactive older adults with mild cognitive impairment (MCI) or mild dementia and to examine how and improve the feasibility and acceptability of the procedures.

ELIGIBILITY:
Inclusion Criteria:

* Age 50+
* Fluent in English
* Diagnosed with MCI or mild dementia
* Physically inactive (< 150 min/wk of planned PA)
* Able to sit in a chair independently for 15+ minutes

Exclusion Criteria:

* Have significant mental or physical disabilities that lead to inability to perform PA safely (e.g., major stroke)
* Severe uncompensated hearing or visual loss
* Having insufficient decisional capacity to consent to participate in research.
* Lack of safety awareness
* Unwilling to be assigned to Pro-Home MeC or control group
* Currently participating in PA intervention research

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2023-03-21 (Actual); Primary Completion 2025-05-05 (Actual); Study Completion 2025-05-05 (Actual)

PRIMARY OUTCOMES:
Program Feasibility | 3 months
  • Program feasibility measured by program adherence (e.g., self-reported program activities in the past 24 hours, yes/no).
Program Acceptability | 3 months
  • Program acceptability measured by patient's perception of the program difficulty. (Too hard, a little too hard, just right, a little too easy, much easy)
Feasibility of NIH Toolbox Cognition Battery | 3 months
  Feasibility of NIH Toolbox Cognition Battery measured by administration time.

SECONDARY OUTCOMES:
NIH Toolbox Cognition Battery scores | 3 months
  NIH Toolbox Cognition Battery Fluid Cognition scores (range 59 - 140, higher score means better cognition)

CONTACTS AND LOCATIONS:
Locations (1):
- Naoko Muramatsu, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No